CLINICAL TRIAL: NCT04239820
Title: Effect of Cladribine Treatment on Microglial Activation in the CNS
Acronym: CLADPET
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 142/2019; 2019-001960-31 (EudraCT Number)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RRMS patients initiating cladribine: Patients will be imaged using PET and MRI at baseline prior the cladribine treatment initiation and 18 months after baseline
  Interventions: Radiation: Imaging

INTERVENTIONS:
Radiation: Imaging — MRI and TSPO-PET imaging at baseline and 18 months after baseline

SUMMARY:
To evaluate the effect of cladribine treatment on microglial activation with conventional MRI, QSM-post processing and TSPO-PET imaging in late stage relapsing remitting multiple sclerosis patients.

DETAILED DESCRIPTION:
Objective: To evaluate with multimodal magnetic resonance (MR) imaging and TSPO-PET imaging whether cladribine treatment has an effect on disease progression-related pathology in late stage relapsing remitting multiple sclerosis (RRMS) patients.

Background: In Multiple Sclerosis (MS), plaques in the white and grey matter of the brain represent the best known pathological changes of the disease, but a significant inflammation process has also been detected outside these plaques in connection with the disease. This extensive, diffuse inflammatory process correlates with the progression of the disease. According to neuropathological research, the diffuse inflammatory process outside the plaques is connected with powerful activation of microglia, oxidative stress, and deficiencies in mitochondrial activity. The activation of microglial cells can be measured in vivo in patients using positron-emission tomography (PET) scanning and so-called 18 kilodalton translocator protein (TSPO) -radioligands. TSPO-radioligands, such as the 11C-PK11195 radioligand, bind to TSPO molecules, which manifest in activated, but not un-activated, microglia.

Cladribine is an immune cell depleting treatment for RRMS. Our hypothesis is that monitoring the treatment of MS could be carried out using TSPO-PET and Quantitative susceptibility mapping (QSM)-MRI scanning, and these multimodal imaging methods could be used to assess the impact of the cladribine medication on the disease process leading to progression and disability by measuring the activation status of microglial cells.

An age-matched historical control group of 10 untreated RRMS patients that have been previously imaged at a 12-18 months interval will be used for comparison.

Study population: 15 late stage RRMS-patients Methods: Clinical evaluation, brain QSM-MRI and PET imaging with 11C-PK11195 radiotracer will be performed at baseline and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent form
* Cladribine treatment is planned and indicated and is according to label
* 45-55 years of age at the time of signing the research informed consent form
* RRMS diagnosis in accordance with McDonald 2017 criteria

Exclusion Criteria:

* Patients with other neurodegenerative disease than MS
* Abnormal lymphocyte counts
* Patients with human immunodeficiency virus (HIV).
* Patients with active chronic infection (tuberculosis or hepatitis).
* Patients with active malignancy.
* Patients with moderate or severe renal impairment (creatinine clearance <60 mL/min)
* Patients that are pregnant or breast-feeding
* Corticosteroid treatment within 4 weeks of imaging
* Patients with significant abnormal findings other than MS in the screening MRI.
* Patients with claustrophobia, or a history of moderate to severe anxiety disorder or panic attacks (which could potentially lead to preterm termination of the imaging)
* Contraindication to PET scan investigations
* Exposure to experimental radiation in the past 12 months such that radiodosimetry limits would be exceeded by participating in this study.
* Intolerance to previous PET scans; i.e. previous hypersensitivity reactions to any PET ligand or imaging agent or failure to participate in and comply with previous PET scans.
* Patients with previous alemtuzumab administration
* Patients with less than 6 months since previous administration of ocrelizumab or rituximab (or with abnormal B-cell counts)
* Patients with less than 1 month since previous administration of other disease modifying therapy

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The research will recruit MS patients who are initiating cladribine treatment and are followed-up at the Neurology Outpatient Clinic at the areas of the Hospital District of Southwest Finland, Helsinki and Uusimaa Hospital District, Pirkanmaa Hospital District and Satakunta Hospital District. The study will not interfere with the initiation or dosage of the medication in any manner. The patient's treating neurologist will select the most suitable medication on the basis of the patient's clinical status, and patients initiating cladribine medication will be offered the option to participate in this imaging study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
11C-PK11195 binding in MS patient brain | baseline, 18 months
  Change in microglia-activity in MS patients during 18 months as measured by 11C-PK11195 PET imaging

SECONDARY OUTCOMES:
MRI metrics | Baseline, 18 months
  To evaluate lesion load of the white matter MS plaques
Expanded Disability Status Scale | Baseline, 18 months
  Expanded Disability Status Scale. The scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Multiple Sclerosis Composite Score | Baseline, 18 months
  Multiple Sclerosis Composite Score which consists of three assessments of walking speed, processing speed and finger dexterity. The scores are combined to provide a Z-score. Lower scores represent greater abnormality.
Blood biomarkers | Baseline, 18 months
  Change in serum neurofilament light (NfL) and glial fibrillary acid protein (GFAP)
11C-PK11195 difference in RRMS and historical healthy controls | Baseline, 18 months
  Difference in microglia-activity between RRMS and historical healthy controls during 18 months as measured by PET imaging and 11C-PK11195
QSM-signal in MS patient brain | baseline, 18 months
  Change in microglia-activity in MS patients during 18 months as measured by QSM-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Laura Airas, Professor, Principal Investigator — Turku University Hospital, division of clinical neurosciences
Locations (1):
- Turku PET Centre, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sjoros T, Saraste M, Matilainen M, Nylund M, Koivumaki M, Kuhle J, Leppert D, Airas L. Serum glial fibrillary acid protein associates with TSPO-expressing lesions in multiple sclerosis brain. Ther Adv Neurol Disord. 2025 Jul 28;18:17562864251352998. doi: 10.1177/17562864251352998. eCollection 2025. PMID 40756531